CLINICAL TRIAL: NCT05803915
Title: Neoadjuvant Toripalimab Plus Nimotuzumab in Primary Limited-Stage Oral Squamous Cell Carcinoma Prior to Radical Therapy：A Single-arm, Phase Ⅱ Study
Brief Title: Neoadjuvant Toripalimab Plus Nimotuzumab in Oral Squamous Cell Carcinoma Prior to Radical Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-ISS-CO407
Record Dates: First submitted 2023-02-28; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-02

CONDITIONS: Oral Squamous Cell Carcinoma
Keywords: Oral Squamous Cell Carcinoma; Toripalimab; Neoadjuvant; PD-1 inhibitor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Toripalimab plus Nimotuzumab (Experimental): The participants will receive 2 doses of neoadjuvant Toripalimab plus Nimotuzumab, then the participants will take a radical surgery or radiotherapy according to the efficacy assessed by investigator per RECIST1.1
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — The participants will receive Toripalimab 240mg intravenous infusion every 3 week, and Nimotuzumab 150mg/㎡ every 2 week for 2 cycles
  Other Names: JS001

SUMMARY:
This study aims to investigate the efficacy and safety of neoadjuvant Toripalimab combined with Nimotuzumab in primary limited stage oral squamous cell carcinoma prior to radical therapy.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the efficacy and safety of neoadjuvant PD-1 inhibitor toripalimab plus nimotuzumab in subjects with primary limited stage, oral squamous cell carcinoma prior to radical therapy. Patients would be treated with neoadjuvant toripalimab plus nimotuzumab for 2 cycles and then received radical surgery or radiotherapy based on the efficacy assessed by investigators per RECIST v1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years old；male or female.
2. Oral squamous cell carcinoma confirmed by cytology or histology. Evaluation by the investigators to confirmed primary limited-stage (clinical stage T1N+M0, T2-4 anyNM0, AJCC 8th) without prior treatment.
3. Patients who are suitable and agree radical therapy.
4. At least 1 evaluable lesion according to RECIST v1.1.
5. ECOG PS ≤ 1
6. Adequate organ function, defined as achieving the following laboratory test results ≤ 14 days before treatment

   1. Patients must meet the following laboratory test results: i. ANC ≥ 1.5 x 10^9 / L ii. Platelets ≥100 x 10^9 / L iii. Hb ≥90 g / L Note: Patients must not receive blood transfusion or growth factor within 14 days before blood sample collection due to neutrophil count, platelet, or hemoglobin below study requirements.
   2. Renal function requirements within 4 weeks before treatment: Endogenous creatinine clearance ≥ 60 mL / min or more (based on 24-hour urine creatinine calculation or Cockcroft-Gault formula method).
   3. Serum total bilirubin ≤ 1.5×ULN (Gilbert syndrome patients can be enrolled if the total bilirubin is <3 × ULN).
   4. AST and ALT ≤ 3 × ULN. If the patient has liver metastases, AST and ALT ≤ 5×ULN
7. Patients with hepatitis B virus (HBV) infection and inactive / asymptomatic HBV carriers; or patients with chronic or active HBV, if HBV DNA <500 IU / mL (or 2500 copies/ mL) will be allowed to enroll. Hepatitis C antibody-positive patients will be allowed to enroll if HCV-RNA is negative during screening.

   NOTE: Patients with detect hepatitis B surface antigen (HBsAg) or HBV DNA, and patients receiving antiviral therapy during screening should be treated for> 2 weeks before enrollment, and Continue treatment for 6 months after study drug therapy
8. Women of childbearing age (WOCBP) must be willing to take effective contraception during the study period and ≥60 days after the last study treatment (including chemotherapy) administration, and the urine or serum pregnancy test result is negative within ≤7 days before treatment.

   a. Women of childbearing age are defined as any woman who has had menarche and has not undergone sterilization (hysterectomy or bilateral ovariectomy) and has not yet reached menopause. Menopause is defined as amenorrhea for 12 months in women> 45 without other biological or physiological causes. In addition, to confirm menopause, women under 55 must have serum follicle stimulating hormone (FSH) levels> 40 mIU / mL.
9. Unsterilized male must be willing to take effective contraception during the study and ≥ 60 days after the last study treatment (including chemotherapy) was administered.

Exclusion Criteria:

1. Not suitable for toripalimab or nimotuzumab treatment.
2. Have previously received any treatment for oral squamous cell carcinoma.
3. Patients with evidence of fistula (esophagus / bronchus or esophagus / aorta)
4. Presence of uncontrollable pleural effusion, pericardial effusion, or ascites that require repeated drainage or medical intervention (with clinically significant recurrence requiring additional intervention within 2 weeks after the intervention).
5. Evidence of complete esophageal obstruction that is not suitable for treatment
6. Have been treated with antitumor agents targeted to PD-1, PD-L1 or PD-L2.
7. Have active meningeal disease or uncontrolled brain metastases.
8. Patients with active autoimmune disease or history of autoimmune diseases may relapse.

   Note: Patients with the following diseases can be entered for further screening:
   1. Controllable type 1 diabetes
   2. Hypothyroidism (only if it could be controlled by hormone replacement therapy)
   3. Controlled celiac disease
   4. Skin diseases that do not require systemic treatment (eg vitiligo, psoriasis, hair loss)
   5. Any other disease that is not expected to recur without external triggers
9. Any active malignancy within ≤ 2 years before treatment, expect specific cancers which being studied in this study and locally recurrent cancers that have been cured (such as resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical cancer and breast cancer in situ).
10. Any condition requiring systemic treatment with corticosteroids (dose above 10 mg / day of prednisone or equivalent dose of similar agents) or other immunosuppressive agents within ≤ 14 days prior to treatment.

    Note: Patients who are currently or previously using any of the following steroid regimens can be enrolled:
    1. Adrenaline replacement (prednisone ≤10mg / day or equivalent dose of similar agents)
    2. Local, ophthalmic, intra-articular, intranasal, and inhaled corticosteroids with minimal systemic absorption.
    3. Prophylactic short-term (≤7 days) use of corticosteroids (for example, to prevent hypersensitivity caused by contrast agent) or to treat non-autoimmune conditions (for example, delayed-type hypersensitivity reactions caused by exposure to allergens).
11. Have a history of interstitial lung disease, non-infectious pneumonia or uncontrolled disease including pulmonary fibrosis, acute lung disease, etc.
12. Severe chronic or active infections (including tuberculosis infections, etc.) that require systemic antibacterial, antifungal, or antiviral treatment within 14 days of treatment.
13. History of HIV infection.
14. Underwent any major surgery requiring general anesthesia ≤ 28 days before treatment.
15. Previously allogeneic stem cell transplantation or organ transplantation.
16. Have any of the following cardiovascular risk factors:

    1. Cardiogenic chest pain occurs within ≤ 28 days prior to treatment and is defined as moderate pain that limits applianceal activities of daily life.
    2. Symptomatic pulmonary embolism occurred within ≤ 28 days before treatment
    3. Acute myocardial infarction occurred within 6 months before treatment
    4. History of heart failure that has reached New York Heart Association Class III or IV ≤ 6 months before treatment.
    5. Ventricular arrhythmia of grade ≥ 2 occurred within ≤ 6 months before treatment
    6. Cerebrovascular accident occurred within ≤ 6 months before treatment
    7. Uncontrolled hypertension: SBP ≥160 mmHg or DBP ≥100 mmHg, although antihypertensive drugs were used ≤ 28 days before treatment or before the first study drug
    8. Any syncope or convulsions ≤ 28 days before treatment
17. History of severe hypersensitivity to other monoclonal antibodies.
18. Have received Chinese herbal medicine or proprietary Chinese medicine for cancer control within 14 days before the first study drug administration.
19. Live vaccinations within ≤ 4 weeks before treatment. Note: Seasonal flu vaccines are usually inactivated vaccines and are allowed. The vaccine used in the nasal cavity is a live vaccine and is not allowed.
20. Presence of basic medical conditions (including abnormal laboratory test values) or alcohol / drug abuse or dependence that are detrimental to study drug administration or affect drug toxicity or AE interpretation, or that may reduce compliance during the study .
21. Participate in another clinical trial at the same time
22. Unintentional weight loss ≥ 5% within 1 month before treatment or severe malnutrition.
23. Nutritional risk index (Shirasu et al 2018) can be used to determine severe malnutrition
24. Pregnant or lactating women
25. Peripheral neuropathy ≥ grade 2 at baseline
26. Uncontrolled diabetes, abnormalities of laboratory tests in potassium, sodium or corrected calcium>grade 1 despite standard medication，or hypoalbuminemia ≥ grade 3 within 14 days before treatment.
27. Have received any chemotherapy, immunotherapy (eg interleukin, interferon, thymosin) or any research treatment within 14 days or 5 half-lives (whichever is longer) before the first study drug administration.
28. Other exclusion criteria

    1. Prisoner or jailer.
    2. People who have been compulsorily detained for the treatment of a mental or physical illness, such as an infectious disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 57 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Major Pathologic response (MPR) rate | up to 18 months
  MPR rate is defined as the proportion of participants who have achieved major pathological response（on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants who have completed the neoadjuvant therapy and underwent surgery.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 18 months
  ORR is defined as the percentage of participants having a complete response or partial response (according to RECIST v1.1) as confirmed by CT or MRI evaluation in all patients who have completed the neoadjuvant therapy.
2-year disease-free survival rate (DFS) | up to 42 months
  DFS is defined as the time from the first day of randomization to the date of first record of disease recurrence or death after radical treatment
2-year progression-free survival rate (PFS) | up to 42 months
  PFS is defined as the time from the first day of randomization to the date of first record of disease progression or death.
2-year overall survival rate (OS) | up to 42 months
  OS is defined as the time from randomization to death due to any cause.
Change in PD-L1 expression | up to 42 months
  Change in the expression of PD-L1 in the tumor tissues from before and after neoadjuvant therapy, based on quantification using immunohistochemistry (IHC) and image analysis.
QoL scores as evaluated by EORTC H&N 35. | up to 42 months
  QoL scores as evaluated the quality of life by EORTC H&N 35.
Incidence and severity of adverse events as evaluated by NCI-CTCAEv5.0. | up to 18 months
  Number of participants experiencing any sign, symptom, disease, or worsening of preexisting conditions associated with the experimental interventions

OTHER OUTCOMES:
Change in Lymphocyte phenotype | up to 42 months
  Changes in the proportion of important immune cells such as CD8+T lymphocytes, CD4+T lymphocytes, dendritic cells (DC) 、NK cells in peripheral blood before and after neoadjuvant therapy, based on quantification using flow cytometry (FCM) and image analysis.
Change in Immunostimulatory cytokines | up to 42 months
  Changes in the proportion of Immunostimulatory cytokines such as Interleukins in peripheral blood before and after neoadjuvant therapy, based on quantification using flow cytometry (FCM) and image analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No